CLINICAL TRIAL: NCT06256133
Title: Impact of Anesthesia-related Enhanced Recovery After Surgery Components on Mortality After Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hyemee Kwon, Assistant professor, Asan Medical Center
Other Study IDs: 2022-0019
Record Dates: First submitted 2024-01-14; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Enhanced Recovery After Surgery; Mortality
Keywords: Pancreaticoduodenectomy; Enhanced Recovery After Surgery; Mortality; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ANS-Surg-ERAS group: fully implementing ERAS pathway including anesthesiology-related components
  Interventions: Procedure: Enhanced Recovery After Surgery protocol
- Surg-ERAS group: preoperative and postoperative ERAS protocol without anesthesiology-related components
- Conventional group: non-ERAS group

INTERVENTIONS:
Procedure: Enhanced Recovery After Surgery protocol — Preoperative oral carbohydrate loading, Ultrasound-assisted thoracic epidural catheter placement, Intraoperative individualized goal-directed fluid therapy, Active warming techniques, The inspired fractional concentration of oxygen was maintained, Multimodal postoperative nausea and vomiting (PONV) prevention strategies, Anesthesia was maintained using a target-controlled infusion (TCI) of propofol and remifentanil, Scheduled administration of an intravenous (IV) or oral nonsteroidal anti-inflammatory drug (NSAID) (50 mg of dexketoprofen)
  Groups: ANS-Surg-ERAS group

SUMMARY:
Pancreaticoduodenectomy (PD), one of the most complex and invasive abdominal surgeries, is associated with long length of stay (LOS) and high morbidity and mortality rates. Enhanced Recovery After Surgery (ERAS) is gaining popularity because it reduces surgical stress and promotes physiological stability through standardized perioperative care, thereby improving the recovery process and outcomes after surgery.

ERAS is a comprehensive approach to perioperative care that involves the collaboration of multiple departments. Within the ERAS program, components primarily implemented by the anesthesiology department include preoperative carbohydrate loading, maintenance of near-zero fluid balance, and multimodal analgesic management, such as midthoracic epidural block. However, they may be underutilized for several reasons, such as deviation from conventional methods (e.g., preoperative carbohydrate loading) or the highly demanding nature of the procedures, which require significant human resources, specialized equipment, and time (e.g., thoracic epidural or transverse abdominis block).

Several randomized trials involving patients undergoing PD have reported that the implementation of ERAS has provided high-level evidence on a safer and quicker recovery, with decreased morbidity rates and shorter LOS than traditional care. Furthermore, a recent study on colorectal surgery reported that the ERAS program may improve not only short-term but also long-term oncological outcomes. However, there is a paucity of research investigating the effects of ERAS on mortality after PD. Furthermore, the impact of anesthesiology-related components within the ERAS pathway has not been extensively studied.

A previously published randomized controlled trial from our institution showed that the outcomes after applying pre- and postoperative ERAS protocols without anesthesiology-related components (Surg-ERAS) were comparable to those of the conventional protocol. This study aimed to compare the short- and long-term mortality rates among patients undergoing PD by examining the same cohort from a previous study, including the conventional (Non-ERAS) and Surg-ERAS groups, in addition to anesthesia fully implementing ERAS programs (ANS-Surg-ERAS group). Moreover, LOS; inflammation parameters, such as neutrophil to lymphocyte ratio (NLR) and C-reactive protein to albumin ratio (CAR); morbidity rate, reoperation rate, and readmission rate were compared among the three groups.

ELIGIBILITY:
* The inclusion cirteria: The participants for this study comprised patients who were enrolled in the previous trial and those who met the same recruitment criteria, except for the inclusion of the ERAS protocol.

  *the previous trial: Hwang DW, Kim HJ, Lee JH, Song KB, Kim MH, Lee SK, Choi KT, Jun IG, Bang JY, Kim SC: Effect of Enhanced Recovery After Surgery program on pancreaticoduodenectomy: a randomized controlled trial. Journal of Hepato-Biliary-Pancreatic Sciences 2019; 26:360-9
* The exclusion criteria were as follows: distant metastasis, recurred periampullary cancer, active or uncontrolled infectious disease, severe psychological or neurological disease, alcohol or drug addiction, overlapping with other clinical trials, pregnancy, uncontrolled cardiopulmonary disease, comorbidities that could affect the quality of life and nutritional status (e.g., liver cirrhosis and renal failure), a history of major abdominal surgery (e.g., gastric resection or colonic resection), the need for simultaneous adjacent organ resection (e.g., portal vein, superior mesenteric vein, transverse colon, and liver), and plan to perform minimally invasive PD.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Department of Hepatobiliary and Pancreatic Surgery initiated the ERAS program without collaborating with the anesthesiology department. Data for 247 patients receiving conventional and Surg-ERAS were extracted from the previous trial from March 2015 to May 2017. Since then, emphasis on the multidisciplinary aspect of the ERAS program has increased, leading to the involvement of the Department of Anesthesiology. From the start of the ERAS collaboration in July 2018, clinical data, including protocol adherence and clinical outcomes, have been prospectively recorded. Subsequently, 355 patients were included and followed up for at least 2 years to assess the relationship between different ERAS bundles and mortality.
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Short- and long-term mortality | 180days and 2years (March 2015 to February 2022)
  The short- (180 days) and long-term (2 years) mortality rates among the three groups

SECONDARY OUTCOMES:
ERAS protocol adherence | Pre-, intraop-, postoperative (during hospitalization) (March 2015 to February 2022)
  Adherance rate of included ERAS protocol components
Length of stay | Postoperative, through study completion (March 2015 to February 2022)
  the number of days from the date of surgery to the date of discharge
Morbidity rate | Within 3 months after surgery (March 2015 to February 2022)
  Postoperative pancreatic fistula (POPF), delayed gastric emptying (DGE), and postpancreatic hemorrhage (PPH), pulmonary complication, acute kidney injury
Re-operation rate | Within 30days after surgery (March 2015 to February 2022)
  Re-operation rate
Re-admission rate | Within 30days after surgery (March 2015 to February 2022)
  Re-admission rate
Inflammatory parameters | On the day before surgery and postoperative day 7 ((March 2015 to February 2022)
  neutrophil-lymphocyte ratio (NLR) and the C-reactive protein (CRP) to albumin ratio (CAR)
Weight change | Pre- and Postoperative(postoperative days 30 and 60) (March 2015 to February 2022)
  comparing the largest difference between baseline body weight before surgery and weight on postoperative days 30 and 60.

CONTACTS AND LOCATIONS:
Overall Officials: Hyemee Kwon, M.D, Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
The dataset used and/or analyzed during the current study is available from the corresponding author upon reasonable request.